CLINICAL TRIAL: NCT05923476
Title: Electroconvulsive Therapy and Concomitant Lithium in Depression: a Double-blind Randomized Controlled Pilot Study
Brief Title: Electroconvulsive Therapy and Concomitant Lithium in Depressive Disorder: A Pilot Study
Acronym: ECT+LITHIUM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC/69072/MH-2021; ID: 2021-03 (Other Grant/Funding Number: Royal Melbourne Hospital)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Lithium and ECT will be administered concomitantly to the intervention group
  Interventions: Drug: Lithium
- Control arm (Placebo Comparator): Placebo and ECT will be administered to the control group
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — Placebo + ECT
  Other Names: Lithicarb

SUMMARY:
Depression is a major psychiatric illness associated with significant morbidity and mortality. Electroconvulsive therapy (ECT) is the most effective treatment for depression and arguably the safest. However, a sizable proportion of patients (20%-30%) do not get well with ECT. Typically, ECT is given as a course extending over weeks and then discontinued. Approximately 50% of patients become unwell again in one year after the completion of ECT even when they use antidepressant medications. Moreover, ECT brings recovery after a series of treatment sessions, usually with a range of 6-20. Each ECT session poses logistic issues. Lithium has robust antidepressant effect when used with antidepressant medications. A combination of lithium and ECT has been studied previously in mania and found to be safe at a lithium level in the human body below 0.6 mEq/L. There is a gap in the literature about the use of lithium and ECT combination in depression. This pilot study aims to investigate the feasibility and safety of conducting a randomized controlled trial comparing lithium and ECT against placebo and ECT. Participants will have either placebo and ECT or lithium ECT at an equal probability. They will be approached for an expression of interest, invited to take part in a consenting session, screened for the eligibility for the study, and assessed for the severity of depression, and cognitive function and then for the improvement in depression. Lithium blood level will be monitored five days after commencement of lithium and each dose change. Participants will be assessed for adverse reactions after each ECT using a formal adverse monitoring report form. Recruitment numbers, trial retention and completion rates and adverse events will be reported.

DETAILED DESCRIPTION:
Title: Electroconvulsive therapy and concomitant lithium in depressive disorder Short Title: ECT and lithium in depression Design: Randomized Controlled Trial-Pilot Study Study Centres: North-Western Mental Health, Hospital: Sunshine Hospital Study Questions: Is a combination of lithium and electroconvulsive therapy (ECT) safe compared with placebo and ECT in patients with a depressive disorder and can this combination be tested in a randomized controlled trial? Study Objectives: To demonstrate the feasibility and safety of conducting a randomized controlled trial of lithium and electroconvulsive therapy against placebo and electroconvulsive therapy.

Inclusion Criteria:

* A depressive episode either in the context of Major Depressive Disorder or bipolar disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, DSM-V, criteria.
* Hamilton Rating Scale for Depression (HRSD 28-item) score of 18 or more.
* Participants who were prescribed ECT as part of standard care.
* Provides written informed consent.

Exclusion Criteria:

* Age below 18 years.
* Contraindication for lithium: renal dysfunction; cardiac disease; concomitant nonsteroidal anti-inflammatory drugs, angiotensin inhibitors and diuretics.
* Neurocognitive disorder (dementia) as defined by DSM-V criteria.
* Serious medical conditions that may preclude ECT or lithium.
* Current or history of non-mood disorder psychosis.
* Pregnancy and lactation based on clinical history and urine pregnancy test.
* A previous history of adverse events to lithium or previous history of lithium toxicity.

Number of Planned Participants:

10 participants in the lithium + ECT group and 10 participants in placebo +ECT group.

Study duration: Two years Investigational product: Lithium

Statistical Methods:

Outcomes Baseline demographic characteristics and variables will be reported with descriptive statistics, mean (SD) or median (25th - 75th percentiles) for continuous variables and frequency (%) for categorical variables.

The number of participants recruited, and their retention rate and the incidence of adverse effects to lithium will be reported. These variables include the severity of depression, the presence of psychotic symptoms, number of previous episodes, the duration of current illness, age, gender, education, socioeconomic status, substance abuse, current medications, and psychiatric and medical comorbidities. Since this is a feasibility study no inferential statistics is planned.

Primary outcome The primary outcome is feasibility as defined as the number of participants who were recruited and randomized and assessed and who received the interventions and remained in the study until completion.

Secondary outcomes

Safety outcomes:

1. Adverse reactions to lithium as defined by

   * Increased rate of post-ECT delirium as measured by time taken for reorientation longer than 30 minutes and defined as DSM-V criteria for delirium.
   * Prolonged seizure, defined as a seizure continuously longer than 120 seconds.
   * Prolonged apnea, defined as apnea longer than 5 minutes.
2. Incidence of lithium toxicity as defined as clinical symptoms and signs which include coarse tremor, disorientation, ataxia (indicating cerebellar involvement) and myoclonus in conjunction with the lithium level above 1.1 mEq/L. If the above symptoms and signs temporally correlated with lithium administration, they will be taken as lithium toxicity even if the lithium level is below 1.1 mEq/L. The study will closely monitor for early warning symptoms and signs, viz., general weakness, diarrhoea, vomiting, a change in the pattern of lithium induced tremor, disorientation and attentional impairment. These early warning symptoms will be treated as lithium manifestations of lithium toxicity in conjunction with a lithium level above 1.1 MeQ/L.
3. Response as defined by 60% reduction or more on HDRS score.

   * The proportion with response (95% CI) will be reported.
   * The speed of remission/response as defined by the number of ECT required. The mean number of treatments (with SD) will be reported.
   * The cognitive outcome, as measured by MoCA and CAMI. The mean scores with SD will be reported.

Since this is a pilot study no inferential statistics is planned. Subgroups: None Consumer Involvement Consumer and carer representatives will provide general support to participants within the scope of their practice. However, they will not be involved in the specific aspects of the study such as recruitment.

ELIGIBILITY:
Inclusion Criteria:

* A depressive episode either in the context of Major Depressive Disorder or bipolar disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, DSM-V, criteria.
* Hamilton Rating Scale for Depression (HRSD 28-item) score of 18 or more.
* Participants who were prescribed ECT as part of standard care.
* Provides written informed consent.

Exclusion Criteria:

* Age below 18 years.
* Contraindication for lithium: renal dysfunction; cardiac disease; concomitant nonsteroidal anti-inflammatory drugs, angiotensin inhibitors and diuretics.
* Neurocognitive disorder (dementia) as defined by DSM-V criteria.
* Serious medical conditions that may preclude ECT or lithium.
* Current or history of non-mood disorder psychosis.
* Pregnancy and lactation based on clinical history and urine pregnancy test.
* A previous history of adverse events to lithium or previous history of lithium toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety | Two years
  Number of participants recruited, retention and completion rate and adverse events

SECONDARY OUTCOMES:
Total ECT sessions | Four weeks
  Number of ECT required
Remission | Four weeks
  Rate of remission
Cognitive function | Four weeks
  Rate of delirium
Relapse of depressive disorder in six months | Six months
  Rate of relapse of depression

CONTACTS AND LOCATIONS:
Overall Officials: A Elias, Principal Investigator — University of Melbourne
Locations (1):
- Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No